CLINICAL TRIAL: NCT02691754
Title: A Cluster Randomised Trial to Measure the Impact of a Free Distribution of Paracetamol to Osteoarthritic Patients on Non-steroidal Anti-inflammatory Drugs (NSAID) and Proton Pump Inhibitors (PPI) Prescription
Brief Title: Impact of a Free Distribution of Paracetamol to Osteoarthritic Patients on Non-steroidal Anti-inflammatory Drugs (NSAID) and Proton Pump Inhibitors (PPI) Prescription
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RePara
Record Dates: First submitted 2016-02-18; First posted 2016-02-25 (Estimated); Last update posted 2025-06-12 (Actual); Status verified 2016-02

CONDITIONS: Osteoarthritis
Keywords: Paracetamol; PPI; Opioids; NSAID; Drug Prescription
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- free paracetamol (Experimental): the General Practitioners can prescribe paracetamol for free (covered by NHS). Patients can receive monthly dose at the local hospital
  Interventions: Other: free paracetamol
- standard drug prescription (No Intervention): Paracetamol is not included in the list of drugs than can be prescribed in charge of National Health System by General Practitioners.
  The General Practitioners can prescribe other drugs or recommend paracetamol payed by the patient (out of pocket) at the chemistry.

INTERVENTIONS:
Other: free paracetamol — General Practitioners can prescribe paracetamol and the patient had to pick up the drug at the local hospital.
  Arms: free paracetamol

SUMMARY:
Paracetamol is recommended as first line treatment for pain control in osteoarthritis, but it is not included in list of drugs than can be prescribed in charge of National Health System by General Practitioners. The hypothesis is that removing this economical barrier the investigators can decrease the prescription of NSAID and of the Proton Pump Inhibitors (PPI), often given for gastric bleeding prophylaxis in NSAID chronic users. As secondary outcome, opioids use was also monitored to see.

Aim of the study is to test if allowing prescription of free paracetamol decreases the prescription of NSAID in osteoarthritic patients.

DETAILED DESCRIPTION:
The trial was conducted in two primary care units of the province of Reggio Emilia. The units have about 34.000 inhabitants. In this units 16 General Practitioners are active, the average beneficiaries per General Practitioner are 1500, about one fourth over 65 years old.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis assisted by a General Practitioners working in Reggio Emilia Province who agreed to participate in the study

Exclusion critera:

- none

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Consumption of NSAID | one year
  Difference in defined daily dose (DDD) per patient between the control and the intervention

SECONDARY OUTCOMES:
Consumption of PPI | one year
  Difference in defined daily dose (DDD) per patient between the control and the intervention
Consumption of opioids | one year
  Difference in defined daily dose (DDD) per patient between the control and the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferretti, MSc, Principal Investigator — Inter-Institutional Pharmaceutical Department, Local Health Authority, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vicentini M, Mancuso P, Giorgi Rossi P, Di Pede S, Pellati M, Gandolfi A, Zoboli D, Ricco D, Busani C, Ferretti A. A cluster randomized trial to measure the impact on nonsteroidal anti-inflammatory drug and proton pump inhibitor prescribing in Italy of distributing cost-free paracetamol to osteoarthritic patients. BMC Fam Pract. 2019 Dec 6;20(1):169. doi: 10.1186/s12875-019-1050-4. PMID 31810456